CLINICAL TRIAL: NCT00527358
Title: Evaluation of SAFER Latinos' Program to Prevent Youth Violence
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Joanne Klevens (U.S. Federal Agency)
Collaborators: George Washington University (Other); Latin American Youth Center (Unknown); Latino Federation of Greater Washington (Unknown)
Responsible Party: Sponsor-Investigator, Joanne Klevens, epidemiologist, Centers for Disease Control and Prevention
Organization: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCIPC-4924
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Violence
Keywords: violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SAFER (Experimental): The intervention community will receive 4 services:
  1. community lay workers will do family outreach and assist families in networking with other families and accessing community services, facilitating parent-youth and family-school communication and homework help for children, and help with translation of school or government/official notices;
  2. youth leaders will provide a supportive presence, help youth navigate the system at school so that they can get help if needed, disseminate information about job training and possibilities, and provide education about avoiding violence;
  3. school support services will offer academic support, acculturation orientation, language, conflict resolution skills training, advocacy and referrals;
  4. Youth drop-in center: will provide youth with an adult supervised place to "hang out", do homework, or participate in sports and job training.
  Interventions: Behavioral: SAFER (Seguridad, Apoyo, Familia, Educacion, y Recursos)
- 2 (No Intervention): Business as usual.

INTERVENTIONS:
Behavioral: SAFER (Seguridad, Apoyo, Familia, Educacion, y Recursos) — 1. community lay workers will do family outreach and assist families in networking with other families and accessing community services, facilitating parent-youth and family-school communication and homework help for children, and help with translation of school or government/official notices;
  2. youth leaders will provide a supportive presence, help youth navigate the system at school so that they can get help if needed, disseminate information about job training and possibilities, provide education about avoiding violence;
  3. school support services will offer academic support, acculturation orientation, language, conflict resolution skills training, advocacy and referrals;
  4. Youth drop-in center will provide youth with an adult supervised place to "hang out", do homework, or participate in sports and job training.
  Arms: SAFER

SUMMARY:
This is an evaluation of a primary prevention program to prevent youth violence by improving family cohesion, networking among families, school bonding, and access to services for Latinos in Langley Park, MD.

DETAILED DESCRIPTION:
To prevent youth involvement in violence, outreach workers will work with families and youth to improve school bonding, family cohesion and awareness and utilization of existing services; and a youth drop-in center will provide youth with an adult supervised place to "hang out", do homework, or participate in sports and job training.

Following implementation of the intervention, we will collect detailed process data (regarding implementation), and evaluate impact/outcome using a quasi-experimental design with baseline (prior to intervention) and two followup data collections in both the intervention and a control community (Culmore, Virginia), measuring change in a selected set of aggregate community variables that represent mediating factors and outcomes for youth violence in Langley Park. Data will be collected via a survey and focus groups.

ELIGIBILITY:
Inclusion Criteria:

* youth 12-24 and their caregiver

Exclusion Criteria:

* residence outside of Langley Park or Culmore

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1400 (Actual)
Dates: Start 2006-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Youth violence | within the next 2 years after intervention started

SECONDARY OUTCOMES:
family cohesion | within the next 2 years after start of intervention
school bonding | within the next 2 years after start of intervention
exposure to antisocial, substance abusing, or violent peers | within the next 2 years after start of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mark Edberg, PhD, Principal Investigator — George Washington University
Locations (1):
- George Washington University, Washington D.C., District of Columbia, United States